CLINICAL TRIAL: NCT06289101
Title: Adapting text4FATHER to Directly Link to First-time Expectant Fathers Using Social Media to Improve Infant and Family Health
Brief Title: text4FATHER R21: Social Media - Efficacy Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); Health Resources and Services Administration (HRSA) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB00422008; R21HD112617 (NIH)
Record Dates: First submitted 2024-02-26; First posted 2024-03-01 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Fathers; Mobile Health; Nuclear Family
Keywords: Fatherhood

STUDY DESIGN:
Intervention Model Description: 2 groups will be enrolled and randomized to receipt or not receipt of the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- text4FATHER (Experimental): Receipt of twice-weekly texts that include resource links and instructions to support behavior change (e.g., videos, infographics) and start mid-pregnancy and continuing through 2 months of baby's age.
  Interventions: Behavioral: text4FATHER
- Usual care (No Intervention): Usual care that is consistent with typical maternity care in involving fathers-to-be.

INTERVENTIONS:
Behavioral: text4FATHER — Receipt of twice-weekly texts that include resource links and instructions to support behavior change (e.g., videos, infographics) and start mid-pregnancy and continuing through 2 months of age.
  Arms: text4FATHER

SUMMARY:
This project will be the first to examine the efficacy of a text messaging intervention designed to recruit first-time fathers-to-be using social media across the U.S. to become involved during pregnancy through two months of postnatal age to support infant, mother, and father well-being.

DETAILED DESCRIPTION:
Father engagement in the prenatal and infant periods is associated with improved infant outcomes (e.g., physical, social and emotional health and development), and mother and father well-being. However, this key window of opportunity has been insufficiently leveraged to promote father engagement, especially, first-time fathers-to-be.

text4FATHER, a multi-modal text messaging program, is designed to increase first-time fathers' knowledge, self-efficacy, and behavioral engagement. text4FATHER sends texts twice-weekly to fathers with threaded content to support infant, partner, and father well-being including resource weblinks to support behavior change from mid-pregnancy through 2 months postnatally. Text content was developed using formative research and feedback from the target population, consensus building with experts, and an evidence-based review.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥18 years
* Live in the U.S.
* Speak English
* Mother gestational age at enrollment less than 25 weeks
* First-time father-to-be
* Willing/able to receive texts.

Exclusion Criteria:

* Individuals who are minors
* Do not speak English
* Unable to provide informed consent
* Not a first-time father
* Not willing/unable to receive texts
* In the past 12 months, any safety concern reported between father-to-be and the mother-to-be, including report of any physical, emotional, sexual harm, threatening behaviors, police involvement, restraining or protective order

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2024-09-10 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Change in Self-efficacy as assessed by the Parenting Sense of Competence Scale (PSOC) | Baseline and 7 months
  Self-report measure with higher score indicating greater confidence in overall parenting skills. This measure is scaled with range from 1 (low) to 6 (high). Mean range 1-6.
Karitane Parenting Confidence Scale (KPCS) | Baseline and 7 months
  Self-report measure with higher score indicating greater confidence in infant care behaviors. This measure is scaled with range from 0 (no, hardly ever) to 3 (yes, most times). Mean range 0-3.
Father Engagement Scale (FES) | Baseline and 7 months
  Self-report measure with higher score indicating greater degree of father engagement in infant care activities. This measure is scaled with range from 0 (never) to 4 (every day or almost every day). Mean range 0-4.

CONTACTS AND LOCATIONS:
Overall Officials: Arik Marcell, MD, MPH, Principal Investigator — Johns Hopkins Dept of Pediatrics / Division of Adolescent/Young Adult Medicine
Locations (1):
- Johns Hopkins University, Baltimore, Maryland, United States

REFERENCES:
- [Background] Marcell AV, Johnson SB, Nelson T, Labrique AB, Eck KV, Skelton S, Aqil A, Gibson D. Protocol for the Feasibility, Acceptability, and Preliminary Efficacy Trial of text4FATHER for Improving Underserved Fathers' Involvement in Infant Care. J Health Care Poor Underserved. 2021;32(3):1110-1135. doi: 10.1353/hpu.2021.0117. PMID 34421016
- [Background] Allport BS, Johnson S, Aqil A, Labrique AB, Nelson T, Kc A, Carabas Y, Marcell AV. Promoting Father Involvement for Child and Family Health. Acad Pediatr. 2018 Sep-Oct;18(7):746-753. doi: 10.1016/j.acap.2018.03.011. Epub 2018 Apr 10. PMID 29653255
- [Background] Allport-Altillo BS, Aqil AR, Nelson T, Johnson SB, Labrique AB, Carabas Y, Marcell AV. Parents' Perspectives on Supporting Father Involvement in African American Families During Pregnancy and Early Infancy. J Natl Med Assoc. 2020 Aug;112(4):344-361. doi: 10.1016/j.jnma.2020.04.002. Epub 2020 May 11. PMID 32409095
- [Background] Aqil A, Allport BS, Johnson SB, Nelson T, Labrique AB, Marcell AV. Content to share with expectant fathers: Views of professionals focused on father involvement. Midwifery. 2019 Mar;70:119-126. doi: 10.1016/j.midw.2018.12.018. Epub 2018 Dec 24. PMID 30611921